CLINICAL TRIAL: NCT01133678
Title: Selection of Chemoradiotherapy Based on Response to Induction Chemotherapy - a Phase II Study in Locally Advanced Squamous Cell Carcinoma of Head and Neck
Brief Title: Study in Locally Advanced Squamous Cell Carcinoma of Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary endpoint reached futility boundary
Sponsor: University of Chicago (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-069-B
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Everolimus; Cisplatin; Paclitaxel; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental): Everolimus 5 mg PO Daily for 2 21-day cycles
  Interventions: Drug: Everolimus
- Placebo (Experimental): Placebo 5 mg PO Daily for 2 21-day cycles
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Phase II Portion (2 21-day cycles of induction therapy) Cisplatin (75 mg/m2 day 1) Paclitaxel (175 mg/m2, day 1) Cetuximab(400 mg/m2 loading dose day 1 then 250mg/m2 weekly ) Everolimus 5 mg PO daily. Following induction patients received [paclitaxel (100 mg/m2 IV weekly), 5-FU (600 mg/m2 IV day 1-5), hydroxyurea 500 mg BID PO (day 1-5), and hyperfractionated twice daily radiotherapy (150 cGy per fraction) day 1-5 of a 14 day cycle which is repeated to deliver the prescribed radiotherapy dose.
  Other Names: Cisplatin, Paclitaxel, Cetuximab, Everolimus
  Arms: Everolimus
Drug: Placebo — Phase II Portion (2 21-day cycles of induction therapy) Cisplatin (75 mg/m2 day 1) Paclitaxel(175 mg/m2, day 1) Cetuximab(400 mg/m2 loading dose day 1 then 250mg/m2 weekly ) Placebo PO daily. Following induction patients received [paclitaxel (100 mg/m2 IV weekly), 5-FU (600 mg/m2 IV day 1-5), hydroxyurea 500 mg BID PO (day 1-5), and hyperfractionated twice daily radiotherapy (150 cGy per fraction) day 1-5 of a 14 day cycle which is repeated to deliver the prescribed radiotherapy dose.
  Other Names: Cisplatin, Paclitaxel, Cetuximab, Placebo
  Arms: Placebo

SUMMARY:
Primary

Compare response rates (relative change in tumor size) to induction chemotherapy consisting of cisplatin/paclitaxel/cetuximab +/- everolimus.

Secondary:

Determine the maximum administered dose (MAD), maximum tolerated dose (MTD), dose limiting toxicity (DLT), and safety of everolimus with cisplatin/paclitaxel/cetuximab induction chemotherapy (phase I portion)

DETAILED DESCRIPTION:
Results reported here are for the randomized, phase II portion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve stage III (hypopharynx, or nasopharynx primary) or stage IVa/IVb (all sites) histologically proven SCCHN with no definitive evidence of metastatic disease
* Patients with unknown primary site of tumor and histologically proven squamous cell carcinoma of a cervical lymph node felt to arise from a site in the head and neck are eligible
* Patients must have at least one measurable site of disease according to RECIST criteria
* Age ≥ 18 years
* Karnofsky performance status > 70%
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Adequate liver function as shown by:
* Serum bilirubin ≤ 1.5 x ULN
* ALT and AST ≤ 2.5x ULN
* INR and PTT ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of randomization.)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients, who have had a major surgery [defined as requiring general anesthesia but not including tonsillectomy, neck dissection, or panendoscopy (triple endoscopy or examination under general anesthesia)], or significant traumatic injury within 4 weeks of start of study drug; patients who have not recovered from the side effects of any major surgery; or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Unequivocal demonstration of metastatic disease (i.e. M1 disease).
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* Severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
* Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* Active (acute or chronic) or uncontrolled severe infections
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Nota bene: subjects that require administration of everolimus through a feeding tube are allowed to participate
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus)
* Patients who have received prior treatment with an mTOR inhibitor for SCCHN (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to everolimus (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* Patients with a know hypersensitivity to cetuximab, cremaphor, paclitaxel, carboplatin, 5FU, hydroxyurea, or any compounds of similar chemical or biologic composition
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Baseline neurologic deficit (> grade II neuropathy)
* Prior severe infusion reaction (grade 4) to a monoclonal antibody

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, M.D., Principal Investigator — The University of Chicago Medical Center
Locations (2):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois

REFERENCES:
- [Derived] Villaflor VM, Melotek JM, Karrison TG, Brisson RJ, Blair EA, Portugal L, De Souza JA, Ginat DT, Stenson KM, Langerman A, Kocherginsky M, Spiotto MT, Hannigan N, Seiwert TY, Cohen EE, Vokes EE, Haraf DJ. Response-adapted volume de-escalation (RAVD) in locally advanced head and neck cancer. Ann Oncol. 2016 May;27(5):908-13. doi: 10.1093/annonc/mdw051. Epub 2016 Feb 15. PMID 26884588
- See also: The University of Chicago Comprehensive Cancer Center Web Page — http://uccrc.uchicago.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Everolimus | Placebo
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 58.1 [42 to 74] | 56.2 [27 to 71] | 57.2 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 21 | 18 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Tumor Responses
Description: Change in tumor size (sum of longest diameters of target lesions) after two cycles of induction therapy, expressed as log of ratio of post-treatment to baseline measure.
Time Frame: Baseline and 2 months
Population: One patient from each arm died prior to cycle 2 and is excluded.
Measure: Mean (Standard Error); unit: dimensionless (log ratio)
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 24 | 24
dimensionless (log ratio) | -0.609 (0.086) | -0.796 (0.112)
Statistical Analysis 1: Comparison: Everolimus vs Placebo; Test type: Other; p = 0.190, t-test, 2 sided — A recommendation to stop the trial early was stipulated if the conditional power at the interim analysis (after 50 patients) was <10% using a stochastic curtailment approach.. This would occur if the interim test statistic is t < -0.287; t-statistic = -1.330, exceeding threshold (<-0.287, conditional power<10%) for early termination

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Everolimus | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 9/25 | 11/25
Other Adverse Events (participants affected / at risk) | 22/25 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=25) | Placebo (N=25)
Alanine aminotransferase increased (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2
Edema limbs (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Fever (General disorders) | 0 | 4
Heart failure (Cardiac disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=25) | Placebo (N=25)
Alanine aminotransferase increased (Infections and infestations) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 8
Anemia (Blood and lymphatic system disorders) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 17 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2
Chills (General disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 15 | 15
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 18 | 20
Diarrhea (Gastrointestinal disorders) | 8 | 9
Dysgeusia (Nervous system disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 6 | 6
Fatigue (General disorders) | 20 | 20
Fever (General disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 5
Lymphocyte count decreased (Investigations) | 0 | 2
Mucosal infection (Infections and infestations) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 20 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 16 | 17
Oral pain (Gastrointestinal disorders) | 11 | 12
Pain (General disorders) | 6 | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 5
Platelet count decreased (Investigations) | 6 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 21 | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 4 | 9
Weight loss (Investigations) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes